CLINICAL TRIAL: NCT06262243
Title: The Effect of Heating With Electrical Blanket After Cesarean Section on the Postpartum Comfort, Pain, Milk Quantity and Breastfeeding Success
Brief Title: The Effect of Heating With Electrical Blanket After Cesarean Section on the Postpartum
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, tuba çıtak, Principal Investigator, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ORDUU-HEM-TÇ-01
Record Dates: First submitted 2024-01-20; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Cesarean Section
Keywords: Caesarean section; electric blanket; nursing

STUDY DESIGN:
Intervention Model Description: The research is a randomized controlled experimental design.
Who Masked: Participant
Masking Description: In this randomized controlled study, 78 mothers, 39 in each group, will be included in the intervention and control groups that meet the criteria for participation in the study. The researcher will give general information about the research to the mothers in the intervention and control groups during hospitalization and nurse admission, and their written informed consent will be obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The group that will receive routine care and electric blankets after cesarean section.
  Interventions: Other: electric blankets
- control group (No Intervention): The group that will receive routine care after cesarean section.

INTERVENTIONS:
Other: electric blankets — While the patient is in surgery; An electric blanket will be placed under the bed mattress, and the bed will be placed on the electric blanket.
  The bed sheet will be laid, and the blanket used in the clinic will be laid on top of the bed sheet.
  -The electric blanket will be turned on at "hot" setting 20 minutes before the patient leaves the surgery. After the mother is placed in a heated bed, the electric blanket will be unplugged when the temperature reaches 36.5.
  Arms: experimental group

SUMMARY:
It is known that maintaining and maintaining normal body temperature in women after cesarean section facilitates the mother's adaptation to the postpartum period. One of the important problems after cesarean section is hypothermia. Therefore, various methods are used to maintain normal body temperature. One of these methods is the use of electric blankets. This study will investigate the effect of using electric blankets after cesarean section on postpartum comfort, pain, milk quantity and breastfeeding success.

DETAILED DESCRIPTION:
After cesarean section, mothers face more problems than mothers who give birth normally. Post-cesarean pain, breastfeeding problems, anesthesia-related side effects, and postpartum complications are important reasons affecting maternal comfort. After a cesarean section, mothers may experience hypothermia due to the low temperature in the operating room, the incision, and the effects of spinal/general anesthesia. In mothers who develop hypothermia after cesarean section, undesirable results may occur in physiological parameters such as fever, pulse, blood pressure, pain, and intestinal motility. Therefore, body temperature, blood pressure, pulse, saturation, pain, time to first flatus and defecation are the main factors that determine patient comfort after surgery. In the postoperative period, both pharmacological and non-pharmacological treatment methods are used to reduce pain, increase the amount of milk, and increase intestinal motility. It is stated in the literature that non-pharmacological methods such as early mobilization, chewing gum, early oral hydration (consumption of water, warm water, tea, coffee), and hot application are effective in increasing intestinal motility. Using active and passive heating methods to prevent hypothermia after cesarean section are practices that affect postpartum comfort. With this study, it is expected that heating with an electric blanket will prevent hypothermia, increase postpartum comfort, reduce pain, and increase breastfeeding success by affecting the amount of milk.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* At least primary school graduate
* The one who is married
* Primiparous women who gave birth at term,
* Having the baby with her after birth
* Those who agreed to participate in the study

Exclusion Criteria:

* Those who gave birth at less than 37 weeks of gestation
* Mothers with babies weighing less than 2500 grams
* The newborn has a congenital anomaly,
* Those with a history of high-risk pregnancy
* Those who received any food, including water, other than breast milk until the 10th day of follow-up
* Those with cardiovascular disease problems, those with a history of neurological diseases
* Mothers with nipple problems
* Diabetes Mellitus, those diagnosed with gestational diabetes mellitus,
* Mothers who gave birth with general anesthesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Postpartum comfort scale | two days
  Postpartum comfort scale, consists of 34 items. A 5-point Likert type scale scoring system was used. For each item, expressions and scoring ranging from "completely agree" (5 points) to "strongly disagree" (1 point) were made. Accordingly, the lowest score to be obtained from the scale is 34 and the highest score is 170.
A Tool to Evaluate the Amount of Breast Milk the Baby Receives | ten days
  It consists of 5 sections: urine amount, breast condition, stool amount, weight and satisfaction, and the features of each section are collected in 3 groups and evaluated out of 0, 1, 2 points. A full score of 10 was considered as the score where breast milk was obtained in the best possible way, and 7 and below were considered as the scores where the breast milk was obtained insufficiently.

SECONDARY OUTCOMES:
Bristol Breastfeeding Assessment Tool | two days
  The scale was developed to evaluate common breastfeeding problems and adequacy in the postpartum period. The mother is observed by the midwife/nurse during breastfeeding, and the mother and baby are evaluated in line with the criteria and a form is filled out. The measurement tool is a Likert-type scale consisting of 4 items: "positioning", "holding", "sucking" and "swallowing".
Insufficient Milk Perception Scale | two days
  The first question asks whether the mother perceives her milk to be sufficient. The mother answers this question with "yes" or "no". Other questions of the scale aim to measure the perception of inadequacy of milk. The mother is asked to score these questions between 0-10. "0" indicates that the milk is perceived as completely inadequate, and "10" indicates that the milk is perceived as completely sufficient. A minimum of 0 and a maximum of 50 points can be obtained from the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru ŞAHİN, Principal Investigator — Ordu Univercity
Locations (1):
- Samsun Training and Research Hospital, Samsun, İ̇lkadim, Turkey (Türkiye)